CLINICAL TRIAL: NCT05230017
Title: Chinese AntiphosPholipid Syndrome cohorT cOllaborative NEtworks
Acronym: CAPSTONE
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jiuliang Zhao, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: 2021-12-28-2.0
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Anti Phospholipid Syndrome
Keywords: anti-phospholipid antibody
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antiphospholipid syndrome (APS) is an autoimmune disorder characterized by thrombosis and pregnancy morbidity in patients with persistently positive antiphospholipid antibodies (aPLs). However, large-scale research on general population with persistent aPLs has been lacking. This project proposes to establish the first multicenter cohort of patients with persistently positive aPLs in China and conduct a comprehensive clinical phenotyping study. Based on traditional phenotypes of thrombotic and pregnancy events, the focus will be on extra-standard clinical phenotypes and prospective assessment of event risk and prognosis in aPL-positive population. A prospective analysis of extra-standard antibodies will also be conducted to recommend detection criteria for extra-standard antibody application in China and to assess their clinical significance.

DETAILED DESCRIPTION:
Chinese AntiphosPholipid Syndrome cohorT cOllaborative NEtworks (CAPSTONE) is a national research network created to register patients with persistent aPLs. We aim at enrolling 2000 patients from a total of six centers, lead by the Peking Union Medical College Hospital (PUMCH). The aPLs assay will be validated in the central lab in PUMCH. All patients will be followed every six months, and up to three years. Thrombotic and pregnancy events related to aPLs will be recorded, as well as extra-criteria clinical phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* The presence of one or more of the antiphospholipid antibodies (aPL) tested according to the 2006 Sapporo APS clasification criteria, on two or more occasions at least 12 weeks apart:

Exclusion Criteria:

* Patients refuse to participate;
* Unable to be followed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with the presense of one or more of the following aPLs can be included, after obtaining the written informed consent. The aPLs include: 1)IgG and/or IgM anticardiolipin antibodies (aCL) in moderate or high titer (>40 GPL or MPL units, respectively, or a titer >99th percentile for the testing laboratory), measured by a standardized enzyme-linked immunosorbent assay (ELISA). 2) IgG and/or IgM anti-beta2-glycoprotein (GP) I >40 GPL or MPL units, respectively, or a titer >99th percentile for the testing laboratory, measured by a standardized ELISA according to recommended procedures. 3) Lupus anticoagulant (LA) activity detected according to published guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular thrombosis related to aPLs | 36 months
  Venous thrombosis, arterial thrombosis, microscopic thrombosis
Pregnancy morbidity related to aPLs | 36 months
  One or more unexplained deaths of a morphologically normal fetus at ≥10 weeks gestation, or one or more premature births of a morphologically normal neonate before 34 weeks gestation because of eclampsia, preeclampsia, or placental insufficiency, or three or more consecutive spontaneous pregnancy losses at <10 weeks gestation, unexplained by chromosomal abnormalities or by maternal anatomic or hormonal causes.

SECONDARY OUTCOMES:
antiphospholipid antibody profile | 36 months
  IgG and/or IgM anticardiolipin (ACL) antibodies, IgG and/or IgM anti-beta2-glycoprotein (GP), Lupus anticoagulant (LA) activity, IgA ACL/anti-β2-GP I，anti-annexin 5 antibody, anti-protein C, anti-protein S, anti-vimentin/cardiolipin complex, and anti-lysobisphosphatidic acid (LBPA) et al.
Extra-criteria manifestations | 36 months
  Thrombocytopenia, haemolytic anemia, APS nephropathy, heart valve lesions, non-stroke CNS manifestations, skin changes (livedo reticularis, leg ulcers)

CONTACTS AND LOCATIONS:
Overall Officials: Jiuliang Zhao, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (18):
- China (18):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affilicated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospical of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University Genral Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No